CLINICAL TRIAL: NCT03297671
Title: Early Identification of Rh Negative Women During Pregnancy and Use of Prophylaxis to Prevent Rh Disease of Newborns in Dadu District, Sindh, Pakistan
Brief Title: The Prevention of Rh Disease of Newborns in Pakistan
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Other Study IDs: Rh Study
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Rhesus Disease; Anti-D (Rh) Antibodies Affecting Care of Mother

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pregnant Women: 2000 pregnant women from the communities in the catchment area of THQ Johi and DHQ Dadu. Rh negative women will receive two RhIg prophylaxis injections.
  Interventions: Drug: RhIg prophylaxis; Device: ELDONCARD; Diagnostic Test: ELDONCARD Test
- Lady Health Visitors (LHVs): 3-5 LHVs who are full time employees at THQ Johi and DHQ Dadu. LHVs will perform ELDONCARD test and provide RhIg prophylaxis injections.
  Interventions: Drug: RhIg prophylaxis; Device: ELDONCARD; Diagnostic Test: ELDONCARD Test

INTERVENTIONS:
Drug: RhIg prophylaxis — Two RhIg prophylaxis injections for Rh negative women
  Other Names: Training on Rh disease
Device: ELDONCARD — ELDONCARD point-of-care test.
Diagnostic Test: ELDONCARD Test — LHVs will perform ELDONCARD test.

SUMMARY:
The investigators aim to demonstrate the feasibility of point-of-care identification of Rh-negative women in a poor, rural setting in Pakistan. Feasibility will be assessed across 2 major domains: 1) acceptance by pregnant women to receive the point-of-care test; and, 2) ability of health workers to administer the point of care test and interpret results. The investigators will also measure whether RhIg prophylaxis can be successfully delivered and is accepted by pregnant women in this setting. The socio-demographic correlates of the acceptance of point-of-care testing and where applicable, the acceptance of RhIg prophylaxis will also be assessed. In addition, the investigators will also explore the baseline knowledge of Rh disease among pregnant women and lady health visitors in this study population and will investigate socio-demographic correlates of baseline knowledge and the uptake of knowledge among pregnant women. Finally, the prevalence of Rh negativity will be calculated and stillbirth and neonatal mortality will be tracked among all participants. All stillbirths and neonatal deaths in this population will be characterized with respect to cause and Rh-negativity.

DETAILED DESCRIPTION:
Rhesus (Rh) disease is a preventable condition caused by an incompatibility between maternal and fetal red blood cells (RBCs). If a person's RBCs lacks a certain protein s/he is said to be Rh-negative. Similarly, if a person's RBCs have that same protein, s/he is said to be Rh-positive. If a pregnant woman's is Rh-negative and her fetus is Rh-positive, the baby is at risk of Rh disease. The complications associated with Rh disease include miscarriage, stillbirth, and neonatal death. Among surviving newborns, Rh disease can cause anemia (low RBCs, which can appear as feeling tired or weak or having a shortness of breath), jaundice (yellowing of the skin), and brain damage. If Rh-negative women are identified, there is a very high chance that Rh disease of the newborn can be prevented.

The purpose of this study is to demonstrate the feasibility of point-of-care identification of Rh-negative women in Dadu district, Pakistan. Determining the Rh status of pregnant women is the first step towards prevention of Rh disease of the newborn. By collecting information about a) the Rh status and blood type of pregnant women; b) the acceptability of a point of care test blood test of Rh disease; and, c) the acceptability of treatment for Rh negativity in pregnant women, the investigators will be able to improve antenatal care and prevent Rh disease of the newborn in rural settings. The implementation of a point-of-care Rh test will allow us for the identification of Rh-negative women, prompt provision of treatment, and prevention of Rh disease of the newborn in rural settings in Pakistan.

As part of this study, participants will be asked a series of questions to assess reproductive history of pregnant women and other demographic characteristics (i.e. questions about home environment and lifestyle). The investigators will also ask whether they are willing to provide a drop of blood, collected via finger prick, to allow us to determine your Rh status by ELDONCARD. If Rh test reveals that the pregnant women are Rh negative, the investigators will offer them up to two doses of treatment, first at approximately 28 weeks of gestation and again within 72 hours of delivery. The injections will be administered at the health facility. They will also be asked to undergo an ultrasound procedure by a trained technician at health facility. Moreover, after the newborn is delivered, the investigators will also ask a series of question and perform an in-person assessment of newborn to assess their health within 72 hours of delivery and then again on their 29th day of life. If they are found to be Rh-negative and they have a miscarriage, stillbirth, or baby dies within the first month of life, the investigators will ask them if we can collect a sample of their blood for further testing.

The investigators will conduct a prospective cohort study in Tehsil Headquarter Hospital (THQ) and District Headquarter Hospital (DHQ) that are situated in Dadu District, Sindh, Pakistan. In total, between 3 and 5 Lady Health Visitors (LHVs) will be enrolled at the study THQ and DHQ to administer the point-of-care test and if necessary, prophylaxis. Over the course of the study period, approximately 2000 pregnant women will be enrolled in total (across both study sites); liveborn newborns delivered to enrolled pregnant women will be followed for the first month of life. The sample size of 2000 pregnant women in this study is driven by the estimated prevalence of Rh negativity in the population (7%) and hence, the number of women investigators expect to offer two injections of RhIg (n=140). A sample size of 140 participants will enable us to measure the acceptance RhIg by pregnant women.

This prospective cohort will include two groups of participants: a) between 3 and 5 LHVs who are full time employees at THQ Johi and DHQ Dadu and, b) 2000 pregnant women from the communities in the catchment area of THQ Johi and DHQ Dadu.

To address one of our study aims, a single questionnaire will be administered to a cadre of approximately 30 health professionals (i.e., physicians, lady health visitors, nurses, etc.) who are not otherwise engaged in study activities.

ELIGIBILITY:
Inclusion criteria for pregnant women

* Pregnant women who present to THQ Johi and DHQ Dadu for ANC
* At least 13 weeks gestation (assessed using self-reported first day of last menstrual period)
* Currently resides within one of 5 Union Council's surrounding THQ Johi and in the catchment area of DHQ Dadu at a fixed address
* Intends to deliver and remain in study catchment area for 1-month after the delivery of their newborn(s)
* Provides written informed consent
* Was not previously enrolled in this study during a different pregnancy

Exclusion criteria for pregnant women

* Previously consented into this study
* Reported that they previously had an anaphylactic reaction to an injection of an antibody blood product
* Has any chronic disease related to the heart, liver, kidney, or lungs
* Does not currently reside within the study's catchment area
* Intends to deliver outside of the catchment area
* Plans to relocate outside of the catchment area within 1-month after the delivery of their newborn(s)
* Does not provide written consent

Inclusion criteria for lady health visitors

* Working full-time at THQ Johi and DHQ Dadu as a Lady Health Visitor
* Verbal consent provided from LHV's direct supervisor
* LHV provides verbal consent to complete a test on baseline knowledge of Rh disease and jaundice
* LHV can attend a 1 day training and orientation session
* LHV provides written informed consent to participate in study

Exclusion criteria for health care workers

* Verbal consent not provided from LHV's direct supervisor
* Does not consent to completing a test on baseline knowledge of Rh disease and jaundice
* Cannot attend a 1 day training and orientation session
* Does not provide written informed consent to participate in study

Non-study health care professional recruitment

A convenience sample of approximately 30 health care professionals including physicians, LHVs, nurses, lady health workers, and midwives, who are not otherwise engaged in study activities will be identified and approached at THQ Johi, DHQ Dadu, and other surrounding health care facilities. To be eligible for participation, health care professionals must not be employed by the study or enrolled in the study as a participant. If health care professionals are determined eligible, they will be asked to complete a short questionnaire to assess their knowledge of Rh disease, similar to the questionnaire administered to LHVs. These health care professionals will not be enrolled into the study or followed prospectively and thus, only verbal consent will be obtained.

Ages: 15 Years to 49 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Study population will be LHVs, pregnant women and non-study health care professional
Sampling Method: Probability Sample
Enrollment: 1654 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of pregnant women who will accept the point of care ELDONCARD test | 12 months
  Acceptability of the point-of-care test will be represented as the proportion of positive (i.e., Yes) responses to each of the 6 questions listed below. The acceptability of the test between sites will be compared.
  1. Did the participant agree to have the point-of-care test?
  2. Do you think that having the point-of-care test will provide information that could improve the health of your newborn?
  3. Do you think the point-of-care test was safe?
  4. Did your family approve of you having the point-of-care test?
  5. Would you recommend the point of care test to other mothers in the village?
  6. In the future, would you agree to have this point of care test again?

SECONDARY OUTCOMES:
Prevalence of Rhesus negativity in pregnant women | 12 months
  Prevalence of Rhesus negativity will be calculated from the total sample size of pregnant women (2000) for the study and the total number of Rhesus-negative women (0-2000) actually identified during the study.
Proportion of lady health visitors who will correctly perform point-of-care test and interpret the results of the point-of-care test | 12 months
  Ability of each lady health visitor to perform point-of-care test, each time a test is performed, a composite score (0-16) will be generated that takes into account all 16 steps of the standardized operational protocol. Composite test scores (0-16) will be plotted over time, where time will be evaluated in increments of days, weeks, and months.
Proportion of positive responses on knowledge pertaining to Rhesus disease in pregnant women and lady health visitors | 12 months
  Knowledge uptake will be assessed in both pregnant women and lady health visitors by comparing their baseline assessments with those completed at the close of the study (proportion of positive (i.e., Yes) responses).
Proportion of pregnant women who will accept RhIg prophylaxis | 12 months
  Acceptability of RhIg prophylaxis will be represented as the proportion of positive (i.e., Yes) responses to each of the 6 questions listed below. The acceptability of RhIg prophylaxis between sites will be compared.
  1. Did the participant verbally agree to receive prophylaxis?
  2. Do you think that receiving prophylaxis may improve the health of your newborn?
  3. Do you think that receiving prophylaxis was safe?
  4. Did your family approve of you receiving prophylaxis?
  5. Would you recommend receiving prophylaxis to other Rhesus-negative mothers in the village?
  6. In future pregnancies, would you agree to receive more injections of RhIg prophylaxis? We will also report the proportion of participants who agreed to receive 1 and/or 2 doses of RhIg in total, and by site.
Rate of stillbirths and neonatal deaths per 1000 live births in this population with respect to cause and Rhesus-negativity | 13 months
  Rate of stillbirths and newborn deaths will be tracked throughout the study and rates will be presented per 1000 live births. Finally, we will also report mean and median antibody titers for all Rhesus-negative women who have a miscarriage, stillbirth, or their newborns die within the first month of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sajid B Soofi, FCPS, Principal Investigator — Aga Khan University; Gul N Khan, MPH, Study Director — Aga Khan University; Shaun Morris, MPH, Principal Investigator — Hospital for Sick-kids Canada; Shabina Ariff, FCPS, Principal Investigator — Aga Khan University; Sidrah Nausheen, FCPS, Principal Investigator — Aga Khan University; Lisa Pell, PhD, Principal Investigator — Hospital for Sick-kids Canada; Alvin Zipursky, MD, Principal Investigator — Eldon Biologicals A/S
Locations (1):
- Taluka Headquarter Hospital Johi and District Headquarter Hospital Dadu, Goth Dado, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Result] Zipursky A, Bhutani VK. Impact of Rhesus disease on the global problem of bilirubin-induced neurologic dysfunction. Semin Fetal Neonatal Med. 2015 Feb;20(1):2-5. doi: 10.1016/j.siny.2014.12.001. Epub 2015 Jan 9. PMID 25582277
- [Result] Fung Kee Fung K, Eason E, Crane J, Armson A, De La Ronde S, Farine D, Keenan-Lindsay L, Leduc L, Reid GJ, Aerde JV, Wilson RD, Davies G, Desilets VA, Summers A, Wyatt P, Young DC; Maternal-Fetal Medicine Committee, Genetics Committee. Prevention of Rh alloimmunization. J Obstet Gynaecol Can. 2003 Sep;25(9):765-73. doi: 10.1016/s1701-2163(16)31006-4. PMID 12970812
- [Result] ELDON K. Simultaneous ABO and Rh groupings on cards in the laboratory or at the bedside. Dan Med Bull. 1955 Mar;2(2):33-40. No abstract available. PMID 14379729
- [Result] Biologicals, E. Clinical Evidence - Comparative Study of EldonCards. 2012
- [Result] Zipursky A, Paul VK. The global burden of Rh disease. Arch Dis Child Fetal Neonatal Ed. 2011 Mar;96(2):F84-5. doi: 10.1136/adc.2009.181172. Epub 2010 Oct 30. No abstract available. PMID 21037283
- [Result] World Health Organization, U., Handbook IMCI. Integrated Management of Childhood Illness. 2005.